CLINICAL TRIAL: NCT04104451
Title: PHASE 1, OPEN-LABEL SAFETY STUDY OF UMBILICAL CORD LINING MESENCHYMAL STEM CELLS (CORLICYTE®) TO HEAL CHRONIC DIABETIC FOOT ULCERS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-1113
Record Dates: First submitted 2019-09-20; First posted 2019-09-26 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 (Experimental)
  Interventions: Drug: Corlicyte
- Dose 2 (Experimental)
  Interventions: Drug: Corlicyte
- Dose 3 (Experimental)
  Interventions: Drug: Corlicyte

INTERVENTIONS:
Drug: Corlicyte — expanded umbilical cord lining mesenchymal stem cells

SUMMARY:
Study Objective:

The objective of this Phase 1 open-label study is to establish the safety and tolerability of Corlicyte mesenchymal stem cells (MSCs) in the treatment of patients with chronic diabetic foot ulcers (DFUs).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Males or non-pregnant, non-lactating females.
2. Age 18 or greater at the time of informed consent.
3. Able and willing to provide written informed consent.
4. Type 1 or Type 2 diabetes.
5. Chronic DFU as the index ulcer meeting all of the following criteria:

   1. present for at least 4 weeks at the time of Screening Visit 1
   2. located below the malleoli of the foot
   3. extends to the dermis or subcutaneous tissue, surrounded by healthy skin, without evidence of exposed muscle, tendon, bone, or joint capsule
   4. area measures 1 to 10 cm2 inclusive, at Screening Visit 1, and
   5. non-healing (defined as ≤50% reduction in ulcer size by the Baseline Visit, as compared to Screening Visit 1).
6. Negative for antibodies to HLA Class I molecules expressed on Corlicyte MSCs, as measured by Luminex HLA single antigen beads, within 3 months prior to start of Treatment Phase without interval sensitizing events.
7. For an index ulcer on the plantar surface of the foot, willingness to offload the foot per study protocol.
8. In women of childbearing potential, willingness to use effective means of birth control during the course of the study; if using systemic birth control, this must have been used for 6 months or longer prior to Screening Visit 1.

Exclusion Criteria:

Exclusion Criteria:

1. Planned DFU treatment to the index ulcer that includes enzymatic agents, cytotoxic agents or any substance(s) that would affect MSC survival during the study period.
2. Women planning to become pregnant during the course of the study.
3. Significant history of, or current evidence of a severe comorbid medical or psychiatric condition such as liver disease, end-stage renal disease, untreated proliferative retinopathy, bleeding diathesis, schizophrenia, or laboratory abnormality that, in the opinion of the Investigator, would preclude enrollment because of unacceptable risk.
4. Presence of any skin condition or skin disorder around the index ulcer that might interfere with the diagnosis of or assessment of study-related endpoints, such as atopic dermatitis, eczema, psoriasis, or seborrheic dermatitis.
5. Presence of actinic keratosis or skin cancer within 2 cm of the index ulcer.
6. Cellulitis or other active infection of the index ulcer or any non-index ulcer at Screening.
7. Use of an investigational agent for ulcer care within 30 days prior to Screening Visit 1.
8. Receipt of an investigational agent or device not approved by the US FDA for marketed use in any indication within 30 days prior to Screening Visit 1.
9. Planned participation in another therapeutic study for any indication prior to completion of study participation.
10. Unwillingness or inability to comply with study visits and study procedures for the entire duration of study participation.
11. Known positivity for Human Immunodeficiency Virus (HIV).
12. Active osteomyelitis or gangrene of either foot at Screening.
13. Known Methicillin-resistant Staphylococcus aureus (MRSA) infection within 30 days prior to Screening Visit 1.
14. Poorly-controlled diabetes mellitus, defined as hemoglobin A1c (HbA1c) >12%.
15. Unsuitable for cellular therapy for any reason, in the opinion of the Investigator.
16. Planned use of cell therapy or amniotic membrane treatment for the index ulcer during study participation.
17. Significant titer of antibodies to HLA Class I molecules expressed on Corlicyte MSCs, as measured by Luminex HLA single antigen beads.
18. Presence of severe peripheral artery disease (PAD) defined as clinical evidence of critical limb ischemia (CLI) during Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
SAE | throughout study completion, an average of 4 months per subject
  Number and percent of subjects in each dosing cohort and overall with a serious adverse reaction to Corlicyte®.

SECONDARY OUTCOMES:
Antibodies to HLA Class I - number and percent | throughout study completion, an average of 4 months per subject
  1. Number and percent of subjects who develop a high titer of antibodies to human leukocyte antigen (HLA) Class I molecules expressed on Corlicyte®
Antibodies to HLA Class I - Time To Development | throughout study completion, an average of 4 months per subject
  2. Time to development of high titer of antibodies to HLA Class I molecules expressed on Corlicyte®
Increase Ulcer Size | throughout study completion, an average of 4 months per subject
  3. Number and percent of subjects with an increase in ulcer size by the end of the Treatment Phase as reviewed by the Wound Core Laboratory (WCL).
Adverse Reaction | throughout study completion, an average of 4 months per subject
  4. Number and percent of subjects with an adverse reaction to Corlicyte® in each cohort and overall.
Suspected Adverse Reaction | throughout study completion, an average of 4 months per subject
  5. Number and percent of subjects with a suspected adverse reaction to Corlicyte® in each cohort and overall.
Suspected Serious Adverse Reaction | throughout study completion, an average of 4 months per subject
  6. Number and percent of subjects with a suspected serious adverse reaction to Corlicyte® in each cohort and overall.
Change in A1c | throughout study completion, an average of 4 months per subject
  7. Change in hemoglobin A1c from Screening to End-of-Study/Early Termination

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Low Wang, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No